CLINICAL TRIAL: NCT02597920
Title: Non-interventional Study Describing Patients' Perception on Anticoagulant Treatment and Treatment Convenience When Treated With Pradaxa or Vitamin K Antagonist for Stroke Prophylaxis in Atrial Fibrillation
Brief Title: Patient Convenience Study
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160.247
Record Dates: First submitted 2015-11-04; First posted 2015-11-05 (Estimated); Results first posted 2019-02-21 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2018-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Switch patients / A: Patients with non-valvular atrial fibrillation (NVAF), currently on Vitamin K Antagonist (VKA) therapy, who are switched to Pradaxa.
- New AF patients / B: Newly diagnosed NVAF patients who are treated with VKA or Pradaxa (VKA : Pradaxa = 1:1).

SUMMARY:
The aim of this non-interventional study is to describe patient's perception of anticoagulant treatment when using Pradaxa® to prevent stroke and systemic embolism while suffering from atrial fibrillation (according to its approved indication in the approved dosages of 110 mg or 150 mg twice daily) in comparison to standard care using Vitamin K Antagonist (VKA).

ELIGIBILITY:
Inclusion criteria:

Cohort A:

1. A. Written informed consent prior to participation
2. A. Female and male patients >= 18 years of age with a diagnosis of non-valvular atrial fibrillation.
3. A. At least 3 months of continuous VKA treatment for stroke prevention prior to baseline assessment.
4. A. Patients switched to Pradaxa® according Summary of Product Characteristics and physician's discretion.

OR

Cohort B:

1. B. Written informed consent prior to participation.
2. B. Female and male patients >= 18 years of age newly diagnosed with non-valvular atrial fibrillation and no previous treatment for stroke prevention (no use of any oral anticoagulant (OAC) within one year prior to enrolment).
3. B. Stroke prevention treatment initiated with Pradaxa® or VKA according to Summary of Product Characteristics and physician's discretion.

Exclusion criteria:

1. Contraindication to the use of Pradaxa® or VKA as described in the Summary of Product Characteristics (SmPC).
2. Patients receiving Pradaxa® or VKA for any other condition than stroke prevention in atrial fibrillation.
3. Current participation in any clinical trial of a drug or device.
4. Current participation in an European registry on the use of oral anticoagulation in AF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: European patients with non valvular atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 1852 (Actual)
Dates: Start 2015-11-11 (Actual); Primary Completion 2017-01-30 (Actual); Study Completion 2017-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (148):
- Belgium (19):
  - 1160.247.1019 Boehringer Ingelheim Investigational Site, Braine-l'Alleud
  - 1160.247.1001 Boehringer Ingelheim Investigational Site, Brussels
  - 1160.247.1018 Boehringer Ingelheim Investigational Site, Brussels
  - 1160.247.1020 Boehringer Ingelheim Investigational Site, Brussels
  - 1160.247.1013 Boehringer Ingelheim Investigational Site, De Pinte
  - 1160.247.1010 Boehringer Ingelheim Investigational Site, Dendermonde
  - 1160.247.1011 Boehringer Ingelheim Investigational Site, Diest
  - 1160.247.1014 Boehringer Ingelheim Investigational Site, Edegem
  - 1160.247.1007 Boehringer Ingelheim Investigational Site, Leuven
  - 1160.247.1021 Boehringer Ingelheim Investigational Site, Lier
  - 1160.247.1002 Boehringer Ingelheim Investigational Site, Maaseik
  - 1160.247.1015 Boehringer Ingelheim Investigational Site, Meise
  - 1160.247.1008 Boehringer Ingelheim Investigational Site, Mol
  - 1160.247.1016 Boehringer Ingelheim Investigational Site, Mol
  - 1160.247.1005 Boehringer Ingelheim Investigational Site, Mons
  - 1160.247.1009 Boehringer Ingelheim Investigational Site, Nijlen
  - 1160.247.1003 Boehringer Ingelheim Investigational Site, Ottignies-Louvain-la-Neuve
  - 1160.247.1012 Boehringer Ingelheim Investigational Site, Roeselare
  - 1160.247.1017 Boehringer Ingelheim Investigational Site, Tienen
- Denmark (8):
  - 1160.247.2006 Boehringer Ingelheim Investigational Site, Frederikssund
  - 1160.247.2008 Boehringer Ingelheim Investigational Site, Herning
  - 1160.247.2001 Sygehus Vendsyssel, Hjørring
  - 1160.247.2007 Hvidovre Hospital, Hvidovre
  - 1160.247.2005 Boehringer Ingelheim Investigational Site, Nykøbing Falster
  - 1160.247.2003 Boehringer Ingelheim Investigational Site, Næstved
  - 1160.247.2009 Boehringer Ingelheim Investigational Site, Roskilde
  - 1160.247.2004 Boehringer Ingelheim Investigational Site, Svendborg
- Greece (72):
  - 1160.247.3410 Boehringer Ingelheim Investigational Site, Agrinio
  - 1160.247.3306 Boehringer Ingelheim Investigational Site, Alexandroupoli
  - 1160.247.3411 Boehringer Ingelheim Investigational Site, Arta
  - 1160.247.3100 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3101 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3102 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3103 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3104 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3105 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3106 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3107 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3108 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3109 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3110 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3111 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3113 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3114 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3116 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3118 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3119 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3120 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3121 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3122 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3200 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3202 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3203 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3204 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3206 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3207 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3208 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3211 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3212 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3213 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3214 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3217 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3218 Boehringer Ingelheim Investigational Site, Athens
  - 1160.247.3316 Boehringer Ingelheim Investigational Site, Chalkidiki
  - 1160.247.3219 Boehringer Ingelheim Investigational Site, Chania
  - 1160.247.3404 Boehringer Ingelheim Investigational Site, Corfu
  - 1160.247.3315 Boehringer Ingelheim Investigational Site, Drama
  - 1160.247.3307 Boehringer Ingelheim Investigational Site, Giannitsá
  - 1160.247.3216 Boehringer Ingelheim Investigational Site, Glyfada, Athens
  - 1160.247.3215 Boehringer Ingelheim Investigational Site, Hrakleion ,Crete
  - 1160.247.3201 Boehringer Ingelheim Investigational Site, Ierapetra, Crete
  - 1160.247.3400 Boehringer Ingelheim Investigational Site, Ioannina
  - 1160.247.3408 Boehringer Ingelheim Investigational Site, Ioannina
  - 1160.247.3409 Boehringer Ingelheim Investigational Site, Ioannina
  - 1160.247.3402 Boehringer Ingelheim Investigational Site, Kalamata
  - 1160.247.3407 Boehringer Ingelheim Investigational Site, Karditsa
  - 1160.247.3318 Boehringer Ingelheim Investigational Site, Katerini
  - 1160.247.3312 Boehringer Ingelheim Investigational Site, Kavala
  - 1160.247.3320 V.Pavlou 21 , Komotini, Komotini
  - 1160.247.3415 Boehringer Ingelheim Investigational Site, Larissa
  - 1160.247.3412 Boehringer Ingelheim Investigational Site, Pátrai
  - 1160.247.3416 Boehringer Ingelheim Investigational Site, Pátrai
  - 1160.247.3317 Boehringer Ingelheim Investigational Site, Serres
  - 1160.247.3300 Boehringer Ingelheim Investigational Site, Thessaloniki
  - 1160.247.3301 Boehringer Ingelheim Investigational Site, Thessaloniki
  - 1160.247.3303 Boehringer Ingelheim Investigational Site, Thessaloniki
  - 1160.247.3304 Boehringer Ingelheim Investigational Site, Thessaloniki
  - 1160.247.3305 Boehringer Ingelheim Investigational Site, Thessaloniki
  - 1160.247.3308 Boehringer Ingelheim Investigational Site, Thessaloniki
  - 1160.247.3309 Boehringer Ingelheim Investigational Site, Thessaloniki
  - 1160.247.3313 Boehringer Ingelheim Investigational Site, Thessaloniki
  - 1160.247.3314 Boehringer Ingelheim Investigational Site, Thessaloniki
  - 1160.247.3319 Boehringer Ingelheim Investigational Site, Thessaloniki
  - 1160.247.3406 Boehringer Ingelheim Investigational Site, Trikala
  - 1160.247.3403 Boehringer Ingelheim Investigational Site, Tripoli
  - 1160.247.3310 Boehringer Ingelheim Investigational Site, Véroia
  - 1160.247.3401 Boehringer Ingelheim Investigational Site, Volos
  - 1160.247.3405 Boehringer Ingelheim Investigational Site, Xánthi
  - 1160.247.3413 Boehringer Ingelheim Investigational Site, Xilokastro
- Netherlands (13):
  - 1160.247.4004 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1160.247.4010 Boehringer Ingelheim Investigational Site, Beugen
  - 1160.247.4013 Boehringer Ingelheim Investigational Site, Capelle aan den IJssel
  - 1160.247.4006 Boehringer Ingelheim Investigational Site, Ede
  - 1160.247.4009 Boehringer Ingelheim Investigational Site, Goes
  - 1160.247.4001 Boehringer Ingelheim Investigational Site, Groningen
  - 1160.247.4008 Boehringer Ingelheim Investigational Site, Heerenveen
  - 1160.247.4012 Boehringer Ingelheim Investigational Site, Heerlen
  - 1160.247.4005 Boehringer Ingelheim Investigational Site, Nijmegen
  - 1160.247.4011 Boehringer Ingelheim Investigational Site, Schiedam
  - 1160.247.4002 Boehringer Ingelheim Investigational Site, The Hague
  - 1160.247.4007 Boehringer Ingelheim Investigational Site, Uden
  - 1160.247.4003 Boehringer Ingelheim Investigational Site, Veldhoven
- Norway (8):
  - 1160.247.5001 Boehringer Ingelheim Investigational Site, Bergen
  - 1160.247.5007 Boehringer Ingelheim Investigational Site, Førde
  - 1160.247.5008 Boehringer Ingelheim Investigational Site, Lierskogen
  - 1160.247.5009 Boehringer Ingelheim Investigational Site, Nesbru
  - 1160.247.5004 Boehringer Ingelheim Investigational Site, Oslo
  - 1160.247.5005 Boehringer Ingelheim Investigational Site, Oslo
  - 1160.247.5010 Boehringer Ingelheim Investigational Site, Stavanger
  - 1160.247.5006 Boehringer Ingelheim Investigational Site, Svelvik
- Portugal (10):
  - 1160.247.6003 Boehringer Ingelheim Investigational Site, Amadora
  - 1160.247.6012 Boehringer Ingelheim Investigational Site, Angra do Heroísmo
  - 1160.247.6007 Boehringer Ingelheim Investigational Site, Aveiro
  - 1160.247.6004 Boehringer Ingelheim Investigational Site, Braga
  - 1160.247.6006 Boehringer Ingelheim Investigational Site, Guimarães
  - 1160.247.6013 Boehringer Ingelheim Investigational Site, Horta
  - 1160.247.6002 Boehringer Ingelheim Investigational Site, Matosinhos Municipality
  - 1160.247.6009 Boehringer Ingelheim Investigational Site, Penafiel
  - 1160.247.6008 Boehringer Ingelheim Investigational Site, Viana do Castelo
  - 1160.247.6005 Boehringer Ingelheim Investigational Site, Vila Franca de Xira
- Sweden (18):
  - 1160.247.7016 Boehringer Ingelheim Investigational Site, Bandhagen
  - 1160.247.7013 Boehringer Ingelheim Investigational Site, Broby
  - 1160.247.7006 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1160.247.7007 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1160.247.7014 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1160.247.7011 Boehringer Ingelheim Investigational Site, Hässleholm
  - 1160.247.7019 Boehringer Ingelheim Investigational Site, Kristianstad
  - 1160.247.7005 Boehringer Ingelheim Investigational Site, Malmo
  - 1160.247.7001 Boehringer Ingelheim Investigational Site, Stockholm
  - 1160.247.7002 Boehringer Ingelheim Investigational Site, Stockholm
  - 1160.247.7003 Boehringer Ingelheim Investigational Site, Stockholm
  - 1160.247.7004 Boehringer Ingelheim Investigational Site, Stockholm
  - 1160.247.7008 Boehringer Ingelheim Investigational Site, Stockholm
  - 1160.247.7010 Boehringer Ingelheim Investigational Site, Stockholm
  - 1160.247.7012 Boehringer Ingelheim Investigational Site, Stockholm
  - 1160.247.7017 Boehringer Ingelheim Investigational Site, Stockholm
  - 1160.247.7009 Boehringer Ingelheim Investigational Site, Värnamo
  - 1160.247.7015 Boehringer Ingelheim Investigational Site, Västerås

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Non-interventional study (NIS) on patients diagnosed with non-valvular atrial fibrillation (NVAF).
Pre-assignment Details: A total of 1852 patients were enrolled, out of which 1822 were found eligible.
Groups:
- Cohort A Pradaxa®: Patients with a diagnosis of non-valvular atrial fibrillation (NVAF), who were using Vitamin K antagonist (VKA) therapy for at least 3 months for stroke prevention before entering the study and were switched to Pradaxa®, received 110 or 150 milligram (mg) twice daily dose of Pradaxa® hard capsules containing Dabigatran etexilate (active ingredient: Dabigatran).
- Cohort B Pradaxa®: Patients newly diagnosed with NVAF, not previously treated with an anticoagulant for the prevention of stroke, and initiated on twice daily dose of 110 or 150 mg Pradaxa® hard capsules containing Dabigatran etexilate (active ingredient: Dabigatran).
- Cohort B VKA: Patients newly diagnosed with NVAF, not previously treated with an anticoagulant for the prevention of stroke, and initiated on VKA therapy. The choice of vitamin K antagonist and the appropriate dosing was at the discretion of the physician.
Period: Overall Study
Arm/Group | Cohort A Pradaxa® | Cohort B Pradaxa® | Cohort B VKA
Started | 585 (Information about study termination is not available for 1 subject.) | 1159 | 78
Completed | 544 | 1075 | 72
Not Completed | 41 | 84 | 6
Not completed — Worsening of other pre-existing disease | 0 | 1 | 0
Not completed — Other adverse event | 20 | 30 | 0
Not completed — Lost to Follow-up | 7 | 9 | 0
Not completed — Refuse to continue in the study | 3 | 13 | 1
Not completed — Other than specified | 10 | 31 | 5
Not completed — Other | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Eligible patients: All patients who took the prescribed treatment and without specific important protocol violations are eligible.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A Pradaxa® | Cohort B Pradaxa® | Cohort B VKA | Total
Number analyzed (Participants) | 585 | 1159 | 78 | 1822
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age (mean and standard deviation (SD)) at the time of signing informed consent form is presented.
  Years | 73.3 (8.9) | 72.7 (9.1) | 74.9 (10.1) | 73.0 (9.1)
Age, Customized [Number; unit: Participants] — Number of participants are presented by age categories.
  Participants
    < 65 years | 83 | 207 | 10 | 300
    ≥ 65 and < 75 years | 213 | 424 | 22 | 659
    ≥ 75 years | 289 | 528 | 46 | 863
Sex: Female, Male [Count of Participants; unit: Participants] — Number of subjects are categorized as Male or Female by each cohort.
  Participants
    Female | 258 | 520 | 43 | 821
    Male | 327 | 639 | 35 | 1001
Race/Ethnicity, Customized [Number; unit: Participants] — Race and ethnicity was not collected under study protocol.
  Participants | NA — Race and ethnicity was not collected under study protocol. | NA — Race and ethnicity was not collected under study protocol. | NA — Race and ethnicity was not collected under study protocol. | NA — Race and ethnicity was not collected under study protocol.
Region of Enrollment [Number; unit: Participants] — Number of subjects are presented by region. Northern European countries included Belgium, Denmark, Norway, Sweden and The Netherlands while the Southern European countries included Greece and Portugal.
  Participants
    Northern Europe | 252 | 447 | 39 | 738
    Southern Europe | 333 | 712 | 39 | 1084
Creatinine clearance at baseline [Number; unit: Participants] — Number of subjects are presented for different categories of creatinine.
  Participants
    <30 milliliter per minute (mL/min) | 0 | 0 | 7 | 7
    30 to < 50 mL/min | 85 | 150 | 23 | 258
    50 to < 80 mL/min | 277 | 510 | 25 | 812
    ≥ 80 mL/min | 168 | 371 | 17 | 556
    Missing | 55 | 128 | 6 | 189
CHA2DS2-VASc stroke risk score at baseline [Number; unit: Participants] — CHA2DS2-VASc score: Congestive heart failure, Hypertension, Age (≥ 75), Diabetes mellitus, Stroke/Transient Ischaemic Attack (TIA), Vascular disease, Age 65-74, Sex category.
  Participants
    Intermediate risk (score = 1) | 48 | 126 | 3 | 177
    High risk (score >=2) | 537 | 1033 | 75 | 1645
HAS-BLED bleeding risk score at baseline [Number; unit: Participants] — HAS-BLED score: Hypertension, Abnormal renal and liver function, Stroke (1 point), Bleeding history or predisposition, Labile International Normalized Ratio (INR), Elderly (>65 years), Drugs and Alcohol.
  Participants
    Low risk (score < 3) | 388 | 1031 | 59 | 1478
    High risk (score >=3) | 197 | 128 | 19 | 344
Speciality of treating physician [Number; unit: Participants] — Number of subjects treated by different physicians are presented
  Participants
    Cardiologist | 548 | 1087 | 67 | 1702
    General practitioner | 23 | 7 | 2 | 32
    Other specialist | 14 | 64 | 8 | 86
    Missing | 0 | 1 | 1 | 2
Type of hospital or practise [Number; unit: Participants] — Number of subjects treated at different type of facilities
  Participants
    Public | 207 | 387 | 33 | 627
    Private | 373 | 753 | 44 | 1170
    Other | 5 | 18 | 0 | 23
    Missing | 0 | 1 | 1 | 2
Owner of medical practice [Number; unit: Participants] — Number of subjects are presented by owner of medical practice
  Participants
    Physician or physician group | 390 | 783 | 39 | 1212
    Health Maintenance Organisation | 7 | 6 | 0 | 13
    Community health center | 24 | 56 | 12 | 92
    Medical / academic health center | 86 | 143 | 13 | 242
    Other hospital | 51 | 140 | 10 | 201
    Other health care corporation | 16 | 8 | 3 | 27
    Other | 11 | 22 | 0 | 33
    Missing | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Perception of Anticoagulant Treatment Questionnaire 2 (PACT-Q2) Scores, for Patients in Cohort A, at Second and Last Assessment Compared to Baseline Assessment
Description: The PACT-Q is a self-administered questionnaire which was developed as a means to investigate patients´ satisfaction with anticoagulant treatment and treatment convenience in patients with deep venous thrombosis (DVT), pulmonary embolism (PE) or atrial fibrillation (AF). The PACT-Q2 is composed of three dimensions covering: convenience (11 items), burden of disease and treatment (2 items), and anticoagulant treatment satisfaction (7 items). Items for convenience and for burden of disease and treatment were reversed (reversed score = 6 - item score), added together and rescaled on a 0-100 scale to obtain the convenience dimension score (CDS). Items for anticoagulant treatment satisfaction are summed and rescaled on a 0-100 scale to determine the satisfaction dimension score (SDS). High scores are more favorable. The two dimension scores are presented for Baseline, Visit 2 (second assessment) and Visit 3 (last assessment) as mean and standard deviation (SD).
Time Frame: Baseline, Visit 2 (7-124 days after initiation on Pradaxa® or VKA), Visit 3 (125-365 days after initiation on Pradaxa® or VKA).
Population: Eligible patients: All patients who took the prescribed treatment and without specific important protocol violations are eligible. PACT-Q2 score obtained after discontinuation of treatment or using incorrect procedure was excluded from the summary for that particular visit.
Measure: Mean (Standard Deviation); unit: Units on Scale
Arm/Group | Cohort A Pradaxa®
Number analyzed (Participants) | 585
Units on Scale
  CDS-Baseline: number analyzed (Participants) | 583
  CDS-Baseline | 63.4 (25.2)
  CDS-Visit 2: number analyzed (Participants) | 567
  CDS-Visit 2 | 77.3 (19.4)
  CDS-Visit 3: number analyzed (Participants) | 543
  CDS-Visit 3 | 79.2 (17.9)
  SDS-Baseline: number analyzed (Participants) | 583
  SDS-Baseline | 53.8 (16.8)
  SDS-Visit 2: number analyzed (Participants) | 567
  SDS-Visit 2 | 67.7 (13.9)
  SDS-Visit 3: number analyzed (Participants) | 543
  SDS-Visit 3 | 70.0 (13.0)
Statistical Analysis 1: Comparison: Cohort A Pradaxa®; Within group comparison of Baseline CDS with that of Visit 2; Test type: Other; p < 0.0001, Paired t-test
Statistical Analysis 2: Comparison: Cohort A Pradaxa®; Within group comparison of Baseline CDS with that of Visit 3; Test type: Other; p < 0.0001, Paired t-test
Statistical Analysis 3: Comparison: Cohort A Pradaxa®; Within group comparison of Baseline SDS with that of Visit 2; Test type: Other; p < 0.0001, Paired t-test
Statistical Analysis 4: Comparison: Cohort A Pradaxa®; Within group comparison of Baseline SDS with that of Visit 3; Test type: Other; p < 0.0001, Paired t-test

2. Primary Outcome: Mean PACT-Q2 Scores, for Patients in Cohort B, at Second and Last Assessment Compared Between Treatment Groups
Description: The PACT-Q2 is composed of three dimensions covering: convenience (11 items), burden of disease and treatment (2 items), and anticoagulant treatment satisfaction (7 items). The PACT-Q2 was to be administered to patients once treatment was ongoing. Items for convenience and for burden of disease and treatment were reversed (reversed score = 6 - item score), added together and rescaled on a 0-100 scale to obtain the convenience dimension score. Items for anticoagulant treatment satisfaction are summed and rescaled on a 0-100 scale to determine the satisfaction dimension score. High scores are more favorable. The two dimension scores are presented for Visit 2 (second assessment) and Visit 3 (last assessment) as mean and standard deviation (SD). Propensity score matching method is used to identify matched Pradaxa® and VKA patients. Only the matched patients in each treatment group are summarized and used for comparison.
Time Frame: Visit 2 (7-124 days after initiation on Pradaxa® or VKA) and Visit 3 (125-365 days after initiation on Pradaxa® or VKA).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on Scale
Arm/Group | Cohort B Pradaxa® | Cohort B VKA
Number analyzed (Participants) | 1159 | 78
Units on Scale
  CDS-Visit 2: number analyzed (Participants) | 63 | 63
  CDS-Visit 2 | 78.3 (13.4) | 69.1 (22.6)
  CDS-Visit 3: number analyzed (Participants) | 62 | 62
  CDS-Visit 3 | 80.3 (10.5) | 69.5 (22.3)
  SDS-Visit 2: number analyzed (Participants) | 63 | 63
  SDS-Visit 2 | 65.9 (7.8) | 58.0 (13.3)
  SDS-Visit 3: number analyzed (Participants) | 62 | 62
  SDS-Visit 3 | 68.4 (8.8) | 58.8 (15.9)
Statistical Analysis 1: Comparison: Cohort B Pradaxa® vs Cohort B VKA; Between group comparison of Visit 2 CDS; Test type: Other; p = 0.0005, Propensity score matching method
Statistical Analysis 2: Comparison: Cohort B Pradaxa® vs Cohort B VKA; Between group comparison of Visit 3 CDS; Test type: Other; p = 0.0002, Propensity score matching method
Statistical Analysis 3: Comparison: Cohort B Pradaxa® vs Cohort B VKA; Between group comparison of Visit 2 SDS; Test type: Other; p = 0.0002, Propensity score matching method
Statistical Analysis 4: Comparison: Cohort B Pradaxa® vs Cohort B VKA; Between group comparison of Visit 3 SDS; Test type: Other; p = 0.0004, Propensity score matching method

3. Primary Outcome: Patient Characterization at Baseline - Categorical Parameters
Description: Categorical parameters of the patient characteristics at baseline included age, gender, Stroke- and/or bleeding related risk factors in medical history and at baseline (MH), co-morbidities (CoMo), concomitant therapies (CM) and dosing of Pradaxa® (DoP).
Time Frame: Baseline
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A Pradaxa® | Cohort B Pradaxa® | Cohort B VKA
Number analyzed (Participants) | 585 | 1159 | 78
Percentage of participants
  Age: < 65 years | 14.2 | 17.9 | 12.8
  Age: ≥ 65 and < 75 years | 36.4 | 36.6 | 28.2
  Age: ≥ 75 years | 49.4 | 45.6 | 59.0
  Gender: Male | 55.9 | 55.1 | 44.9
  Gender: Female | 44.1 | 44.9 | 55.1
  MH: Thromboembolism | 14.0 | 9.1 | 12.8
  MH: Cardiovascular Conditions | 22.4 | 18.5 | 21.8
  MH: Bleedings | 4.1 | 2.5 | 7.7
  MH: Other Conditions | 8.2 | 6.4 | 9.0
  CoMo: Thromboembolism | 5.8 | 4.0 | 9.0
  CoMo: Cardiovascular Conditions | 79.7 | 79.4 | 82.1
  CoMo: Bleedings | 3.6 | 2.6 | 7.7
  CoMo: Other Conditions | 21.9 | 18.4 | 25.6
  CM: Antihypertensives | 84.8 | 81.1 | 84.6
  CM: Lipid modifying agents | 45.3 | 42.6 | 51.3
  CM: Antiarrhythmic agents | 29.4 | 25.4 | 19.2
  CM: Proton pump inhibitors | 18.8 | 15.9 | 26.9
  CM: Antithrombotic agents | 7.4 | 10.1 | 21.8
  CM: Amiodarone | 3.9 | 5.0 | 2.6
  CM: Antidepressants | 4.4 | 4.3 | 6.4
  CM: Verapamil | 3.6 | 2.8 | 1.3
  CM: H2-receptor antagonists | 2.1 | 0.9 | 0.0
  CM: NSAIDS | 0.5 | 1.1 | 2.6
  DoP: 110 mg twice daily: number analyzed (Participants) | 585 | 1159 | 0
  DoP: 110 mg twice daily | 55.9 | 57.3 |
  DoP: 150 mg twice daily: number analyzed (Participants) | 585 | 1159 | 0
  DoP: 150 mg twice daily | 44.1 | 42.7 |

4. Primary Outcome: Patient Characteristics at Baseline - CHA2DS2-VASc Stroke Risk Score and HAS-BLED Bleeding Risk Score
Description: CHA2DS2-VASc stroke risk score is calculated based on the following conditions: Congestive heart failure, Hypertension, Age (≥ 75), Diabetes Mellitus, Stroke/ Transient Ischaemic Attack (TIA), Vascular disease, Age 65-74, Sex category. HAS-BLED bleeding risk score is calculated based on the following conditions: Hypertension, Abnormal renal and Hypertension, Abnormal renal and liver function, Stroke (1 point), Bleeding history or predisposition, Labile INR, Elderly (>65 years), Drugs and Alcohol. CHA2DS2-VASc stroke risk score may range from 0 to 9 with 0 being the best outcome. HAS-BLED bleeding risk score may range from 0 to 9 with 0 being the best outcome. CHA2DS2-VASc stroke risk score and HAS-BLED bleeding risk score at baseline are patient characteristics.
Time Frame: Baseline
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Cohort A Pradaxa® | Cohort B Pradaxa® | Cohort B VKA
Number analyzed (Participants) | 585 | 1159 | 78
Units on scale
  CHA2DS2-VASc | 3.4 (1.5) | 3.2 (1.4) | 3.8 (1.3)
  HAS-BLED | 2.1 (0.9) | 1.7 (0.8) | 2.0 (1.0)

5. Primary Outcome: Patient Characterization at Baseline - Creatinine Clearance
Description: Creatinine clearance at baseline is a measure of the patient's kidney function and is one of the baseline patient characteristics.
Time Frame: Baseline
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: millilitre/ minute [mL/min]
Arm/Group | Cohort A Pradaxa® | Cohort B Pradaxa® | Cohort B VKA
Number analyzed (Participants) | 585 | 1159 | 78
millilitre/ minute [mL/min] | 74.40 (27.08) | 75.89 (26.60) | 63.83 (37.55)

6. Primary Outcome: Patient Characteristics at Baseline - Vitamin K Antagonist Treatment Duration
Description: Vitamin K Antagonist (VKA) treatment duration at baseline is only applicable for Cohort A patients and is one of the baseline patient characteristics.
Time Frame: Baseline
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Cohort A Pradaxa® | Cohort B Pradaxa® | Cohort B VKA
Number analyzed (Participants) | 585 | 0 | 0
Years | 4.44 (3.65) |  |

7. Secondary Outcome: Mean PACT-Q2 Scores, for Patients in Cohort A, at Last Assessment Compared to Second Assessment
Description: The PACT-Q2 is composed of three dimensions covering: convenience (11 items), burden of disease and treatment (2 items), and anticoagulant treatment satisfaction (7 items). The PACT-Q2 was to be administered to patients once treatment was ongoing. Items for convenience and for burden of disease and treatment were reversed (reversed score = 6 - item score), added together and rescaled on a 0-100 scale to obtain the convenience dimension score. Items for anticoagulant treatment satisfaction are summed and rescaled on a 0-100 scale to determine the satisfaction dimension score. High scores are more favorable. The two dimension scores are presented for Visit 2 (second assessment) and Visit 3 (last assessment) as mean and standard deviation (SD).
Time Frame: Visit 2 (7-124 days after initiation on Pradaxa® or VKA) and Visit 3 (125-365 days after initiation on Pradaxa® or VKA).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on Scale
Arm/Group | Cohort A Pradaxa®
Number analyzed (Participants) | 585
Units on Scale
  CDS-Visit 2: number analyzed (Participants) | 567
  CDS-Visit 2 | 77.3 (19.4)
  CDS-Visit 3: number analyzed (Participants) | 543
  CDS-Visit 3 | 79.2 (17.9)
  SDS-Visit 2: number analyzed (Participants) | 567
  SDS-Visit 2 | 67.7 (13.9)
  SDS-Visit 3: number analyzed (Participants) | 543
  SDS-Visit 3 | 70.0 (13.0)
Statistical Analysis 1: Comparison: Cohort A Pradaxa®; Within group comparison of Visit 2 CDS with that of Visit 3; Test type: Other; p < 0.0001, Paired t-test
Statistical Analysis 2: Comparison: Cohort A Pradaxa®; Within group comparison of Visit 2 SDS with that of Visit 3; Test type: Other; p < 0.0001, Paired t-test

8. Secondary Outcome: Description of PACT-Q1 Items for Patients in Cohort B at Baseline
Description: The PACT-Q1 is composed of a single dimension (7 items), covering the expectations of patients regarding their anticoagulant treatment, and was to be administered before treatment initiation. The 7 items are: A1: How confident are you that your anticoagulant treatment will prevent blood clots? A2: Do you expect that your anticoagulant treatment will relieve some of the symptoms you experience? A3: Do you expect that your anticoagulant treatment will cause side effects such as minor bruises or bleeding? A4: How important is it for you to have an anticoagulant treatment that is easy to take? A5: How concerned are you about making mistakes when taking your anticoagulant treatment? A6: How important is it for you to take care of your anticoagulant treatment by yourself? A7: How concerned are you about how much you pay for your anticoagulant treatment? Responses ranged from 1 (Not at all) to 5 (Extremely/ Completely/ Very much).
Time Frame: Baseline
Population: Eligible patients: All patients who took the prescribed treatment and without specific important protocol violations are eligible. PACT-Q1 score at Visit 1 obtained after discontinuation of treatment or using incorrect procedure was excluded from the summary.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Cohort B Pradaxa® | Cohort B VKA
Number analyzed (Participants) | 1148 | 77
Units on scale
  A1: number analyzed (Participants) | 1147 | 77
  A1 | 3.8 (0.8) | 3.7 (0.8)
  A2: number analyzed (Participants) | 1146 | 77
  A2 | 3.1 (1.2) | 2.8 (1.2)
  A3: number analyzed (Participants) | 1147 | 77
  A3 | 2.7 (0.9) | 2.8 (1.0)
  A4: number analyzed (Participants) | 1147 | 77
  A4 | 4.2 (0.8) | 3.8 (1.0)
  A5: number analyzed (Participants) | 1147 | 77
  A5 | 2.8 (1.4) | 2.9 (1.4)
  A6: number analyzed (Participants) | 1147 | 77
  A6 | 4.1 (0.9) | 3.9 (1.0)
  A7: number analyzed (Participants) | 1147 | 77
  A7 | 2.9 (1.4) | 2.8 (1.5)

ADVERSE EVENTS:
Time Frame: From signing the informed consent till end of the study; up to 290 days
Description: In this non-interventional study the analysis of Adverse Events (AE) was based on collected serious or non-serious Adverse Drug Reactions (ADR) and fatal Adverse Events for eligible patients only.
Arm/Group | Cohort A Pradaxa® | Cohort B Pradaxa® | Cohort B VKA
All-Cause Mortality (participants affected / at risk) | 1/585 | 5/1159 | 1/78
Serious Adverse Events (participants affected / at risk) | 4/585 | 8/1159 | 2/78
Other Adverse Events (participants affected / at risk) | 0/585 | 0/1159 | 0/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A Pradaxa® (N=585) | Cohort B Pradaxa® (N=1159) | Cohort B VKA (N=78)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Lung adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
This study was conducted in an unblinded manner so site and patient selection bias could have occurred. Therefore, current practice patterns at these sites may not necessarily reflect patterns of care elsewhere.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2015-07-17): https://cdn.clinicaltrials.gov/large-docs/20/NCT02597920/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT02597920/SAP_001.pdf